CLINICAL TRIAL: NCT03929211
Title: A Phase I/II Study of CPI-613 and Hydroxychloroquine for Patients With High Risk MDS Who Have Failed Hypomethylating Therapy
Brief Title: CPI-613 and Hydroxychloroquine for Patients With High Risk Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administrative withdrawal by IRB
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057945; WFBCCC 99119 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH); NCI-2019-02787 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Myelodysplastic Syndromes; Progressive Disease
Keywords: Relapsed/refractory myelodysplastic syndrome; Failed hypomethylating therapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Disease Progression | interventions — devimistat; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 and hydroxychloroquine (Experimental): The initial phase of the study will be a dose escalation of hydroxychloroquine from 600 mg to 1,200 mg orally flat dose given 2 hours before the CPI-613 infusion on days 1-5 of every 28 days. CPI-dose will be 2,000 mg/m² and will not be escalated.
  Interventions: Drug: CPI-613; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: CPI-613 — Given intravenously, CPI-613 dose will be 2,000 mg/m² and will not escalate.
  Other Names: 6,8-Bis(benzylthio)octanoic Acid
Drug: Hydroxychloroquine — Given by mouth, hydroxychloroquine will be dose escalated from 600 mg to 1,200 mg orally given 2 hours before the CPI-613 infusion on days 1-5 of every 28 day cycle in a 3+3 dose escalation design.
  Other Names: 118-42-3, hydroxychloroquine, HYDROXYCHLOROQUINE, Hydroxychloroquine

SUMMARY:
This is a phase 1/2 study of the combination of CPI-613 and hydroxychloroquine for the treatment of high risk myelodysplastic syndrome patients who have failed a hypomethylating agent.

DETAILED DESCRIPTION:
Primary Objective(s):

* To determine the Maximum Tolerated Dose (MTD) of the combination of CPI-613 and Hydroxychloroquine therapy for patients with high risk MDS who have failed hypomethylating therapy.
* To determine the overall response rate (complete remission (CR), marrow CR, partial remission (PR), Hematologic improvement (HI)) of high risk MDS patients who have failed hypomethylating agents, treated with the combination of CPI-613 and the maximally tolerated dose of hydroxychloroquine

Secondary Objective(s):

* To assess the safety of the combination
* To assess progression-free-survival (PFS)
* To assess the overall survival of MDS patients who have failed hypomethylating agents treated with the combination of CPI-613 and hydroxychloroquine defined as the time from enrolment on study to death from any cause.
* To assess any changes in the frequency of blood transfusions

OUTLINE: This is a phase I, dose-escalation study of hydroxychloroquine, followed by a phase II study.

Patients receive hydroxychloroquine orally (PO) and 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-5. Treatments repeat every 14 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 3, patients receive hydroxychloroquine PO and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria before enrollment:

* Histologically documented high risk MDS whose disease has failed to respond, progressed or relapsed while on a hypomethylating agent.
* IPSS-R score of Intermediate, high or very high at time of enrollment
* ECOG Performance Status of ≤3.
* Men and women 18 years of age or older.
* Expected survival >2 months.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* Patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities. Patients with persisting, non-hematologic, non-infectious toxicities from prior treatment ≤ Grade 2 are eligible, but must be documented as such.
* Laboratory values obtained ≤2 weeks prior to enrollment must demonstrate adequate hepatic function, renal function, and coagulation as defined below:
* Aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL]
* Alanine aminotransferase [ALT/SGPT] ≤3x UNL
* Bilirubin ≤1.5x UNL
* Serum creatinine ≤1.5 mg/dL or 133 μmol/L
* Albumin ≥ 2.0 g/dL or ≥ 20 g/L.
* Mentally competent, ability to understand and willingness to sign an IRB-approved written informed consent form.
* Have access via central line (e.g., portacath).

Exclusion Criteria:

* Patients with the following characteristics are excluded:
* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, symptomatic coronary artery disease, myocardial infarction within the past 3 months, uncontrolled cardiac arrhythmia, pericardial disease or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.
* Patients with active central nervous system (CNS) or epidural tumor.
* Any active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any condition or abnormality which may, in the opinion of the investigator, compromise his or her safety.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Lactating females.
* Life expectancy less than 2 months.
* Unwilling or unable to follow protocol requirements.
* Evidence of ongoing uncontrolled serious infection.
* Requirement for immediate palliative treatment of any kind including surgery.
* Patients with uncontrolled HIV infection. (Note: Patients with known HIV infection are excluded because patients with an immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, and because there may be unknown or dangerous drug interactions between CPI-613 and anti-retroviral agents used to treat HIV infections).
* Patients who have received radiotherapy, surgery, treatment with cytotoxic agents (except a hypomethylating agent, i.e. azacytidine or decitabine), treatment with biologic agents, immunotherapy, or any other anti-cancer therapy of any kind, or any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of CPI-613 treatment.
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities | 4 weeks
  Dose-limiting toxicities assessed in order to be able to establish the maximum tolerable dose for the combination of CPI-613 and Hydroxychloroquine therapy for patients with high risk myelodysplastic syndrome who have failed hypomethylating therapy. Using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for adverse event reporting (Grade 1 (Mild) - 5 (Death) as well as expectedness (unexpected/expected) and attribution (definitely related to study treatment to unrelated to study treatment).
Overall Response Rate | 4 weeks
  Measurements for response criteria will be based upon the Modified International Working Group (IWG) 2006 response criteria for altering natural history of myelodysplastic syndrome. Overall response rates criteria - complete remission (CR), partial response (PR) marrow CR, hematologic improvement (HI), or stable disease, failure, relapse after complete response or partial response, cytogenetic response, disease progression and survival) of high risk myelodysplastic syndrome patients who have failed hypomethylating agents treated with the combination of CPI-613 and the maximally tolerated dose of hydroxychloroquine.

SECONDARY OUTCOMES:
Proportion of Patients with Toxicities | 4 weeks
  Toxicity profiles of participants during the trial to assess the safety of the combination of CPI-613 and hydroxychloroquine will be presented in tables that describe the number and proportion of patients observed with toxicities.
Progression-free-survival | Up to 5 years or until death
  Progression-free-survival is defined as the duration of time from the start of treatment to the time of progression, death, or date of last contact; those lost to follow-up will be censored. Kaplan-Meier survival curves to examine progression free survival in participants will be created.
Overall Survival | Up to 5 years or until death
  Overall survival of myelodysplastic syndrome patients who have failed hypomethylating agents treated with the combination of CPI-613 and hydroxychloroquine defined as the time from enrollment on study to death from any cause.
Changes in the Frequency of Blood Transfusions | Baseline to approximately 6 months
  The investigators will assess for each participant the number of blood transfusions needed and create tables to display the number and timing of blood transfusions that occur.

CONTACTS AND LOCATIONS:
Overall Officials: Bayard Powell, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No